CLINICAL TRIAL: NCT05953636
Title: The Effect of Different Timings of Protein Supplementation on Variable Outcomes in Hemodialysis Patients
Brief Title: Effect of Different Timings of Protein Supplementation in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Timing of protein in HD
Record Dates: First submitted 2023-07-01; First posted 2023-07-20 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Protein Supplementation
Keywords: Timing; Protein Supplementation; hemodialysis

STUDY DESIGN:
Intervention Model Description: This research is a randomized multi-center clinical trial in which 120 hemodialysis patients will be randomly assigned to one of the study groups.
  * Group A: 40 patients will receive oral protein nutritional supplement (ONS) (Fresubin protein powder 25mg/5scoops per hemodialysis session) for 8 weeks 1 hour before the start of the session (pre-dialytic).
  * Group B: 40 patients will receive oral protein nutritional supplement (ONS) for 8 weeks 2 hours after the start of the session (intra-dialytic).
  * Group C: 40 patients will receive oral protein nutritional supplement (ONS) for 8 weeks in non-dialysis days (inter-dialytic).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pre-dialytic (Other): 40 patients will receive oral protein nutritional supplement (ONS) (Fresubin protein powder 25mg/5scoops per hemodialysis session) for 8 weeks 1 hour before the start of the session (pre-dialytic).
  Interventions: Dietary Supplement: oral protein nutritional supplement (ONS) (Fresubin protein powder 25mg/5scoops per hemodialysis session)
- intra-dialytic (Other): 40 patients will receive oral protein nutritional supplement (ONS) for 8 weeks 2 hours after the start of the session (intra-dialytic).
  Interventions: Dietary Supplement: oral protein nutritional supplement (ONS) (Fresubin protein powder 25mg/5scoops per hemodialysis session)
- inter-dialytic (Other): 40 patients will receive oral protein nutritional supplement (ONS) for 8 weeks in non-dialysis days (inter-dialytic).
  Interventions: Dietary Supplement: oral protein nutritional supplement (ONS) (Fresubin protein powder 25mg/5scoops per hemodialysis session)

INTERVENTIONS:
Dietary Supplement: oral protein nutritional supplement (ONS) (Fresubin protein powder 25mg/5scoops per hemodialysis session) — oral protein nutritional supplement (ONS) (Fresubin protein powder 25mg/5scoops per hemodialysis session) given in group A (predialytic: 1 hour before the start of the session), in group B (intradialytic: 2 hours after the start of the session ), in group C (interdialytic: in non-dialysis days )

SUMMARY:
The aim of this work is to study the effect of different timings of protein supplementation on variable outcomes in hemodialysis patients.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a prevalent chronic condition and the incidence of end-stage renal disease (ESRD) is expected to increase over the next few decades. In patients with CKD, especially in those with ESRD and undergoing maintenance dialysis therapy (MDT), a state of metabolic and nutritional derangements, more aptly called protein-energy wasting (PEW), caused by a combination of insufficient intake, uremic toxins, inflammation, and superimposed catabolism, plays a major role among the many risk factors that affect outcomes of CKD. PEW, showing a high prevalence (up to 50-75%) in patients with CKD stages 4-5, is closely associated with both increased morbidity/mortality risk and worsens quality of life.

Oral nutritional supplement (ONS) is a simple and effective way to supplement energy and protein to malnourished patients on the basis of regular diet. Therefore, if the protein of regular diet in dialysis patients are not enough, they should be supplemented with (ONS) when appropriate.

It is common for nephrologists to prescribe oral nutritional supplements (ONS), but the compliance to these at prescribed doses is relatively low. While directly administering ONS during hemodialysis (HD) ensures compliance and has been shown to improve nutritional status in these patients, the risks of intradialytic hypotension, inadequate dialysis, hygiene issues, and staff burden remain major deterrents for caregivers from formulating policies with regard to intradialytic meals.

ELIGIBILITY:
Inclusion Criteria:

* Adult hemodialysis patients (≥18 years of age).
* Received dialysis for at least 6 months prior to study screening.
* Receive hemodialysis at least 3 times per week .

Exclusion Criteria:

* Receiving nutritional supplementation prior to study commencing or within 1 month of commencement in the study .
* Participants with an allergy to any ingredients in the nutritional supplements.
* Significant edema and fluid overload.
* Hepatic patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
effect on nutritional status | 6 weeks
  assessment of nutritional status change at 6 weeks from baseline using Subjective Global Assessment (SGA)
effect on blood pressure | 6 weeks
  systolic and diastolic Blood pressure change at 6 weeks from baseline
effect on dialysis adequacy | 6 weeks
  Estimation of Kt/V change at 6 weeks from baseline

SECONDARY OUTCOMES:
effect on BMI | 6 weeks
  BMI assessment change at 6 weeks from baseline
effect on serum albumin | 6 weeks
  • serum albumin change at 6 weeks from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mamdouh Elsayed, MD, Principal Investigator — lecturer; Amr Mohamed El Kazaz, MBBCh, Study Chair — resident
Locations (1):
- Faculty of Medicine, Aexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kalantar-Zadeh K, Ikizler TA, Block G, Avram MM, Kopple JD. Malnutrition-inflammation complex syndrome in dialysis patients: causes and consequences. Am J Kidney Dis. 2003 Nov;42(5):864-81. doi: 10.1016/j.ajkd.2003.07.016. PMID 14582032
- [Background] Carrero JJ, Nakashima A, Qureshi AR, Lindholm B, Heimburger O, Barany P, Stenvinkel P. Protein-energy wasting modifies the association of ghrelin with inflammation, leptin, and mortality in hemodialysis patients. Kidney Int. 2011 Apr;79(7):749-56. doi: 10.1038/ki.2010.487. Epub 2010 Dec 22. PMID 21178976
- [Background] Ikizler TA, Cano NJ, Franch H, Fouque D, Himmelfarb J, Kalantar-Zadeh K, Kuhlmann MK, Stenvinkel P, TerWee P, Teta D, Wang AY, Wanner C; International Society of Renal Nutrition and Metabolism. Prevention and treatment of protein energy wasting in chronic kidney disease patients: a consensus statement by the International Society of Renal Nutrition and Metabolism. Kidney Int. 2013 Dec;84(6):1096-107. doi: 10.1038/ki.2013.147. Epub 2013 May 22. PMID 23698226
- [Background] Agarwal R, Georgianos P. Feeding during dialysis-risks and uncertainties. Nephrol Dial Transplant. 2018 Jun 1;33(6):917-922. doi: 10.1093/ndt/gfx195. PMID 28633456
- [Background] Kistler BM, Benner D, Burrowes JD, Campbell KL, Fouque D, Garibotto G, Kopple JD, Kovesdy CP, Rhee CM, Steiber A, Stenvinkel P, Ter Wee P, Teta D, Wang AYM, Kalantar-Zadeh K. Eating During Hemodialysis Treatment: A Consensus Statement From the International Society of Renal Nutrition and Metabolism. J Ren Nutr. 2018 Jan;28(1):4-12. doi: 10.1053/j.jrn.2017.10.003. PMID 29249295
- [Derived] Elsayed MM, Elkazaz AM. The effect of different timings of protein supplementation on variable outcomes in hemodialysis patients: a randomized clinical trial. Clin Exp Nephrol. 2025 May;29(5):672-680. doi: 10.1007/s10157-025-02626-7. Epub 2025 Jan 18. PMID 39826005